CLINICAL TRIAL: NCT07299500
Title: Retrospective Descriptive Study of a Cohort of Non-HIV Immunocompromised Patients With Toxoplasmosis at the Strasbourg University Hospital From 2010 to 2023
Brief Title: Study of a Cohort of Non-HIV Immunocompromised Patients With Toxoplasmosis at the Strasbourg University Hospital
Acronym: TOXO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9375
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Toxoplasmosis
Keywords: Cerebral toxoplasmosis; HIV; Immunodeficiencies; Hematopoietic stem; stem cell transplantation
MeSH Terms: conditions — Toxoplasmosis, Cerebral; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Toxoplasmosis in HIV-positive individuals is well-studied and has a codified management protocol, which is not the case for other immunodeficiencies, except for recent recommendations in the context of hematopoietic stem cell transplantation. A description of this population is necessary to estimate the number of patients affected and to define their specific management (diagnosis, treatment, prevention).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Immunocompromised (i.e., solid organ transplant recipient, hematological malignancy, cancer patient, patient treated with immunosuppressive therapy or therapy affecting the immune system by any mechanism, hematopoietic stem cell transplant recipient, patient with an autoimmune disease or immunodeficiency, whether primary or secondary).
* At least one positive toxoplasmosis PCR test (regardless of tissue)

Exclusion Criteria:

* Subject who has expressed opposition to the reuse of their data for scientific research.
* HIV positive
* Congenital toxoplasmosis
* Isolated ocular toxoplasmosis in immunocompetent individuals

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥18 years) with a positive toxoplasmosis PCR test (regardless of tissue)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Overall patient survival rates | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'immunologie clinique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France